CLINICAL TRIAL: NCT04351750
Title: Dose-response of Physical Exercise on Pelvic Floor Muscle Function in Postmenopausal Women With Urinary Incontinence: a Randomized Controlled Trial
Brief Title: Dose-response of Physical Exercise on Pelvic Floor Muscle Function in Postmenopausal Women With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kuan-Yin Lin, Assistant professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-108-091
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-06

CONDITIONS: Urinary Incontinence; Pelvic Floor Muscle Weakness
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-intensity group (Experimental): The participants will receive high-intensity general exercise and pelvic floor muscle training in high-intensity group. The intensity of aerobic exercise is 60 ~ 89% of heart rate reserve (HRR) or oxygen uptake reserve (VO2R), which is equivalent to the vigorous intensity exercise proposed in the American College of Sports Medicine (ACSM). The intensity of resistance exercise is 60~80% of 1 repetition maximum (RM), which is equivalent to the moderate-to-vigorous intensity exercise proposed in ACSM. After finishing the general exercise, participants will receive pelvic floor muscle training.
  Interventions: Other: general exercise; Other: pelvic floor muscle training
- low-intensity group (Experimental): The participants will receive low-intensity general exercise and pelvic floor muscle training in low-intensity group. The intensity of aerobic exercise is 40~59% of HRR or VO2R, which is equivalent to the moderate intensity exercise proposed in ACSM. The intensity of resistance exercise is 40~50% of 1RM, which is equivalent to the very light-to-light intensity exercise proposed in ACSM. After finishing the general exercise, participants will receive pelvic floor muscle training.
  Interventions: Other: general exercise; Other: pelvic floor muscle training
- control group (Active Comparator): The participants will only receive pelvic floor muscle training in control group.
  Interventions: Other: pelvic floor muscle training

INTERVENTIONS:
Other: general exercise — The participants will receive training sessions twice a week for 8 weeks. General exercise includes aerobic exercise (stationary bike) and resistance training (thera-band, sandbags, dumbbell and swiss ball), and the intensity and progression of both aerobic and resistance exercises will be provided as recommended by the ACSM, and the exercise will individualized based on participant's HRR, 1 RM weight and Borg Scale of Perceived Exertion Scale (Borg RPE scale). An oximeter will be utilized to monitor the heart rate and SPO2 of the participants to ensure safety during the training session.
  Arms: high-intensity group; low-intensity group
Other: pelvic floor muscle training — Participants will do pelvic floor muscle training in different positions. Each session includes three sets of eight to twelve maximum voluntary contractions of pelvic floor muscle, with holding the contraction for 6 to 8 seconds, and if possible, to do three fast contractions at the end of each set.

SUMMARY:
Urinary incontinence (UI) symptoms are highly prevalent among women, and menopause is one of the risk factors for UI. During the menopausal transition, not only the hormonal secretion is changed but also the level of physical activity is affected. The time spent on physical activity is reduced in postmenopausal women. Studies have shown that physical activity acts in a bidirectional manner, exerting either a preventive or an aggravating effect on urinary incontinence. Individuals with sedentary lifestyle and insufficient physical activity (< 150 min/week) are at risk of developing UI, and regular physical activity exerts a protective effect in preventing UI, but the optimal type, duration, and intensity of exercise for the female older adult population remain unknown. In addition, objective measurements of pelvic floor muscle function is needed as the use of self-reported measures may cause response bias. The aim of the study is to investigate the effect of different intensity of exercise on pelvic floor muscle function and HRQoL in postmenopausal women with UI. The investigators hypothesize that (a) both high- and low-intensity physical activities can improve pelvic floor muscle strength and HRQoL in postmenopausal women with UI, and (b) the improvement in high-intensity group is higher than that in low-intensity group. A randomized trial will be conducted to compare the effect of different exercise intensity on pelvic floor muscle function in postmenopausal women with urinary incontinence (n=90).

DETAILED DESCRIPTION:
In Taiwan, the prevalence of urinary incontinence (UI) in postmenopausal women was 29.8%. Previous studies have indicated that menopause may be associated with developing UI. As there are many estrogen receptors in pelvic floor, the estrogen decline after menopausal transition may lead to pelvic floor muscle dysfunction, and the subsequent development of UI. Pelvic floor muscle training (PFMT) has been recommended by the International Continence Society as the first-line conservative treatment for women with UI. In addition to the prevalent incontinence associated with postmenopausal status, many women tend to have a more sedentary lifestyle after menopausal transition. Previous studies have shown that a sedentary lifestyle is related to UI in older women and indicated the importance of physical activity on preventing incontinence. Regular physical exercise including aerobic exercise and resistance training has been proved to improve bone mineral density, stress management and autonomic functions in postmenopausal women. However, the effect of different intensity of physical exercise adding to PFMT on pelvic floor muscle function in postmenopausal women with UI remains unknown. Therefore, the aim of this study is to investigate the effect of different intensity of exercise on pelvic floor muscle function and health-related quality of life in postmenopausal women with UI.

This is a randomized controlled trial (RCT). Postmenopausal women with UI and a sedentary lifestyle will be recruited. Eligible participants will be randomly allocated to the high-intensity group to receive high intensity general exercise plus PFMT program, the low-intensity group to receive low intensity general exercise plus PFMT, or the control group to receive only PFMT. The intervention will be provided twice weekly for eight weeks. The assessments will be conducted at baseline and after 8-week intervention. The primary outcome is pelvic floor muscle function measured by manometry and through digital palpation. The secondary outcomes are symptom severity measured using the International Consultation on Incontinence Questionnaire -Urinary Incontinence Short Form (ICIQ-UI SF), health-related quality of life measured using the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol), and physical activity levels measured by the International Physical Activity Questionnaire (IPAQ). In addition, the participants will be asked to complete a 3-day bladder diary. Data analysis will be performed using Statistical Product and Service Solutions (SPSS) version 22.0. For continuous data, analysis of covariance tests will be used for within-group and between-group comparisons, respectively. For categorical data, McNemar's tests and chi-square tests will be used for within-group and between-group comparisons. The significant level is set at p-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women: amenorrhoea for longer than 12 months.
* Symptomatic UI: The questionnaire for urinary incontinence diagnosis (QUID) score >0
* Sedentary lifestyle: < 150 minutes of moderate-intensity aerobic physical activity throughout the week, or < 75 minutes of vigorous-intensity aerobic physical activity throughout the week, or an equivalent combination of moderate and vigorous-intensity activity
* Able to answer the questionnaire correctly (no language barrier or cognitive problems)
* No other physical or psychological problem that would interfere participation in the study
* No concurrent outpatient rehab attendance / supervised exercise

Exclusion Criteria:

* Use hormone therapy
* Age >80 y/o
* Neurological condition: Spinal cord injury, multiple sclerosis, transverse myelitis, cerebrovascular accident
* Radical surgery for pelvis, sling, and prolapse surgery
* Malignancy for bladder, urethra, uterus, ovary, cervix, and rectum
* Overflow incontinence or voiding dysfunction

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Yin Lin, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nygaard I, Shaw J, Egger MJ. Exploring the association between lifetime physical activity and pelvic floor disorders: study and design challenges. Contemp Clin Trials. 2012 Jul;33(4):819-27. doi: 10.1016/j.cct.2012.04.001. Epub 2012 Apr 12. PMID 22521947
- [Background] Bo K, Nygaard IE. Is Physical Activity Good or Bad for the Female Pelvic Floor? A Narrative Review. Sports Med. 2020 Mar;50(3):471-484. doi: 10.1007/s40279-019-01243-1. PMID 31820378
- [Background] Faleiro DJA, Menezes EC, Capeletto E, Fank F, Porto RM, Mazo GZ. Association of Physical Activity With Urinary Incontinence in Older Women: A Systematic Review. J Aging Phys Act. 2019 Dec 1;27(4):906-913. doi: 10.1123/japa.2018-0313. PMID 30859902
- [Background] Akkus Y, Pinar G. Evaluation of the prevalence, type, severity, and risk factors of urinary incontinence and its impact on quality of life among women in Turkey. Int Urogynecol J. 2016 Jun;27(6):887-93. doi: 10.1007/s00192-015-2904-5. Epub 2015 Dec 5. PMID 26638154
- [Background] Duval K, Prud'homme D, Rabasa-Lhoret R, Strychar I, Brochu M, Lavoie JM, Doucet E. Effects of the menopausal transition on energy expenditure: a MONET Group Study. Eur J Clin Nutr. 2013 Apr;67(4):407-11. doi: 10.1038/ejcn.2013.33. Epub 2013 Feb 20. PMID 23422924
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Barry MJ, Fowler FJ Jr, O'leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT; Measurement Committee of the American Urological Association. The American Urological Association Symptom Index for Benign Prostatic Hyperplasia. J Urol. 2017 Feb;197(2S):S189-S197. doi: 10.1016/j.juro.2016.10.071. Epub 2016 Dec 22. PMID 28012747
- [Background] Kelleher CJ, Cardozo LD, Khullar V, Salvatore S. A new questionnaire to assess the quality of life of urinary incontinent women. Br J Obstet Gynaecol. 1997 Dec;104(12):1374-9. doi: 10.1111/j.1471-0528.1997.tb11006.x. PMID 9422015
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Li YT, Tsai YJ, Wang LY, Ou YC, Kao YL, Lin KY. The feasibility of a multimodal exercise program for sedentary postmenopausal women with urinary incontinence: A pilot randomized controlled trial. Maturitas. 2023 Jan;167:90-98. doi: 10.1016/j.maturitas.2022.10.004. Epub 2022 Oct 27. PMID 36327627
- See also: What are pelvic floor safe exercises? — http://www.pelvicfloorfirst.org.au/pages/pelvic-floor-safe-resistance-exercises.html
- See also: International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form — https://iciq.net/iciq-ui-sf
- See also: International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module — https://iciq.net/iciq-lutsqol

RESULTS

PARTICIPANT FLOW:
Groups:
- High-intensity Group: The participants will receive high-intensity general exercise and pelvic floor muscle training in high-intensity group. The intensity of aerobic exercise is 60 ~ 89% of heart rate reserve (HRR), which is equivalent to the vigorous intensity exercise proposed in the American College of Sports Medicine (ACSM). The intensity of resistance exercise is 60~80% of 1 repetition maximum (RM), which is equivalent to the moderate-to-vigorous intensity exercise proposed in ACSM. After finishing the general exercise, participants will receive pelvic floor muscle training.
  general exercise: The participants will receive training sessions twice a week for 8 weeks. General exercise includes aerobic exercise (stationary bike) and resistance training (thera-band, sandbags, dumbbell and swiss ball), and the intensity and progression of both aerobic and resistance exercises will be provided as recommended by the ACSM, and the exercise will individualized based on participant's HRR, 1 RM weight and Borg Scale of Perceived Exertion Scale. An oximeter will be utilized to monitor the heart rate and SPO2 of the participants to ensure safety during the training session.
  pelvic floor muscle training: Participants will do pelvic floor muscle training in different positions. Each session includes three sets of eight to twelve maximum voluntary contractions of pelvic floor muscle, with holding the contraction for 6 to 8 seconds, and if possible, to do three fast contractions at the end of each set.
- Low-intensity Group: The participants will receive low-intensity general exercise and pelvic floor muscle training in low-intensity group. The intensity of aerobic exercise is 40~59% of HRR, which is equivalent to the moderate intensity exercise proposed in ACSM. The intensity of resistance exercise is 40~50% of 1RM, which is equivalent to the very light-to-light intensity exercise proposed in ACSM. After finishing the general exercise, participants will receive pelvic floor muscle training.
  general exercise: The participants will receive training sessions twice a week for 8 weeks. General exercise includes aerobic exercise (stationary bike) and resistance training (thera-band, sandbags, dumbbell and swiss ball), and the intensity and progression of both aerobic and resistance exercises will be provided as recommended by the ACSM, and the exercise will individualized based on participant's HRR, 1 RM weight and Borg Scale of Perceived Exertion Scale. An oximeter will be utilized to monitor the heart rate and SPO2 of the participants to ensure safety during the training session.
  pelvic floor muscle training: Participants will do pelvic floor muscle training in different positions. Each session includes three sets of eight to twelve maximum voluntary contractions of pelvic floor muscle, with holding the contraction for 6 to 8 seconds, and if possible, to do three fast contractions at the end of each set.
Period: Overall Study
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
Started | 14 | 15 | 18
Completed | 12 | 13 | 13
Not Completed | 2 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-intensity Group | Low-intensity Group | Control Group | Total
Number analyzed (Participants) | 12 | 13 | 13 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (6.1) | 65.6 (8.63) | 62.3 (8.8) | 64.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 13 | 38
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 12 | 13 | 13 | 38
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Weight (kg)/Height (m) squared
  kg/m^2 | 24.06 (4.52) | 25.44 (5.64) | 24.95 (4.92) | 24.75 (4.92)

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Floor Muscle Function Measured by Digital Palpation
Description: Pelvic floor muscle function (muscle strength) was measured through digital palpation. Three times of maximum contraction holding for five seconds with an interval resting of five seconds were performed, and the maximum value among three was recorded as the muscle strength of maximal voluntary contraction (MVC). The result was recorded using the modified Oxford grading scale, a six-point system with higher score indicated stronger muscle strength (0 = no contraction, 1 = flicker, 2 = weak, 3 = moderate with lift, 4 = good with lift, 5 = strong with lift).
Time Frame: absolute values at 8 weeks
Population: There were three missing data of pelvic floor muscle function (high-intensity group n=1, low-intensity group n=1, control group n=1) as the participants declined the assessment due to embarrassment with the test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
Number analyzed (Participants) | 11 | 12 | 12
score on a scale | 4.00 (0.89) | 3.25 (0.87) | 3.75 (1.14)

2. Primary Outcome: Pelvic Floor Muscle Function Measured by Manometry
Description: The manometry supplied by Laborie® Biofeedback and Stimulation System was used to assess vaginal squeeze pressure, and the unit of pressure was registered in millimeter of mercury (mmHg). The participants were asked to perform 3 times of MVC, holding for 5 seconds with 5 seconds interval resting time, and the maximum value among the three MVC was recorded. The muscle strength was calculated as the value of MVC minus resting tone.
Time Frame: absolute values at 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
Number analyzed (Participants) | 11 | 12 | 12
mmHg | 16.64 (21.55) | 8.58 (7.64) | 13.23 (13.92)

3. Secondary Outcome: International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form
Description: The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form will be used to assess the severity of UI symptoms. The total score ranges from 0 to 21; a higher score indicates greater severity.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
Number analyzed (Participants) | 12 | 13 | 13
score on a scale | 6.75 (3.62) | 4.92 (3.67) | 7.15 (4.28)

4. Secondary Outcome: International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life
Description: The International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life will be used to evaluate quality of life in UI patients. The total score ranges from 19 to 76. A higher score indicates greater impact on quality of life.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
Number analyzed (Participants) | 12 | 13 | 13
score on a scale | 32.17 (9.46) | 27.85 (8.76) | 32.69 (7.01)

5. Secondary Outcome: International Prostate Symptom Score
Description: The International Prostate Symptom Score will be used to evaluate the severity of lower urinary tract symptoms. The total score ranges from 0 to 35. A higher score indicates greater severity.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
Number analyzed (Participants) | 12 | 13 | 13
score on a scale | 7.25 (3.62) | 6.31 (4.89) | 8.23 (5.88)

6. Secondary Outcome: 3-day Bladder Diary
Description: The participants had to record the frequency of daytime urination for three days but not necessarily consecutive. Daytime frequency was defined as the number of voids since first void after waking to last void before sleep.
Time Frame: absolute values at 8 weeks
Population: There were four missing data in total (high-intensity group n=1, low-intensity group n=1, control group n=2) as the participants did not return the diary or the recording information was incomplete.
Measure: Mean (Standard Deviation); unit: voids per day
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
Number analyzed (Participants) | 11 | 12 | 11
voids per day | 7.76 (1.21) | 8.00 (2.64) | 8.18 (2.24)

7. Secondary Outcome: International Physical Activity Questionnaire
Description: The International Physical Activity Questionnaire will be used to measure participants' physical activity levels. The questionnaire assessed the time people spending in physical activity in the last seven days, and the intensity of physical activity level was divided into vigorous, moderate, and walking. The total physical activity levels were calculated by a formula: total MET-minutes/week (Metabolic equivalent of task- minutes per week) = Vigorous intensity (8.0 METs*min*day) + Moderate intensity (4.0 METs*min*days) + Walking (3.3 METs*min*days). A higher score indicates a greater physical activity levels.
Time Frame: absolute values at 8 weeks
Population: There were two missing data of physical activity levels (low-intensity group n=1, control group n=1) as the participants reported "not sure" in the time spending in physical activity.
Measure: Mean (Standard Deviation); unit: MET-min/week
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
Number analyzed (Participants) | 12 | 12 | 12
MET-min/week | 2624.35 (1390.43) | 2133.54 (1024.29) | 1814.25 (1511.58)

ADVERSE EVENTS:
Time Frame: through 8 week intervention
Arm/Group | High-intensity Group | Low-intensity Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT04351750/Prot_SAP_000.pdf